CLINICAL TRIAL: NCT02247115
Title: Rapid Assessment of Trainee Endoscopy Skills (RATES) Study: A Prospective Multicenter Study Evaluating Competence in Endoscopic Ultrasound and Endoscopic Retrograde Cholangiopancreatogram Among Advanced Endoscopy Trainees
Brief Title: Rapid Assessment of Trainee Endoscopy Skills (RATES) Study
Acronym: RATES
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Brigham and Women's Hospital (Other); Carolinas Medical Center (Other); Columbia University (Other); Dartmouth-Hitchcock Medical Center (Other); Virginia Mason Hospital/Medical Center (Other); Geisinger Clinic (Other); Henry Ford Hospital (Other); Indiana University (Other); Johns Hopkins University (Other); Mayo Clinic (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Icahn School of Medicine at Mount Sinai (Other); New York Presbyterian Brooklyn Methodist Hospital (Other); Northwestern University Feinberg School of Medicine (Other); The University of Texas Health Science Center, Houston (Other); University Hospitals Cleveland Medical Center (Other); Fox Chase Cancer Center (Other); University of California, Los Angeles (Other); University of Kansas Medical Center (Other); University of Texas (Other); University of Virginia (Other); University of Wisconsin, Madison (Other); Vanderbilt University Medical Center (Other); Washington University School of Medicine (Other); Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0604
Record Dates: First submitted 2014-09-15; First posted 2014-09-23 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Competency-Based Education
Keywords: endoscopic ultrasound; endoscopic retrograde cholangiopancreatography; competency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The establishment of a number of training programs in therapeutic endoscopy, standardization of the performance of endoscopic ultrasound (EUS) and endoscopy retrograde cholangiopancreatography (ERCP) and definition of competence is of paramount importance. The length of training and minimum number of procedures, requisite theoretical learning and methodology to define competence in EUS and ERCP are not well defined. The investigators research has demonstrated that individuals in training acquire skills at different rates and the number of procedures completed alone is a suboptimal marker for competency in a given procedure. Hence, emphasis needs to be shifted away from the number of procedures performed to performance metrics with well-defined and validated thresholds of performance. Multicenter prospective data are needed to help guide development of competency based medical education that define learning curves in EUS and ERCP and set evidence-based benchmarks required to achieve competence using a validated competency assessment tool.

Hypothesis: The central hypothesis is that a validated EUS and ERCP competency assessment tool will allow for reliable and generalizable standardized learning curves, competency benchmarks and creation of a centralized national database that compares a trainee's performance amongst peers.

DETAILED DESCRIPTION:
Competency-based medical education and milestones: Given the increasing emphasis on quality metrics and competency in health care, the Accreditation Council for Graduate Medical Education (ACGME) recently announced plans to replace their current reporting system in 2014 with the Next Accreditation System (NAS). This reporting system focused on: 1) ensuring that milestones are reached at various points in training, 2) ensuring that competence is achieved by all trainees, and 3) making certain that these assessments are documented by their programs.

Learning curves and competence in EUS: EUS is a vital tool in the diagnosis and staging of gastrointestinal and certain non-gastrointestinal malignancies and diseases. EUS is operator dependent and training in EUS requires the development of technical and cognitive skills beyond that required for standard endoscopic procedures. It is intuitive that the quality of EUS in provision of patient care is directly proportional to the training, skill and experience of the endosonographer. Unfortunately, the intensity and length of training and minimum number of procedures required, requisite curriculum and extent of theoretical learning, and methodology to define competence are not well defined. There are limited data on learning curves in EUS imaging. Based on expert opinion, the ACGME recommends a minimum of 150 total supervised procedures, 75 of which have a pancreatobiliary indication and 50 cases of fine needle aspiration (FNA) (25 of which are pancreatic FNA) before competency can be determined.

Similar guidelines were recently proposed by the British Society of Gastroenterology (BSG) and the European Society of Gastrointestinal Endoscopy. However, these guidelines have not been validated. This does not account for the different rates at which people learn and in fact, many experts believe that the majority of trainees will require double the number of proposed procedures to achieve competency in EUS.

Learning curves and competence in ERCP: ERCP is an effective modality in the evaluation and management of pancreatobiliary diseases. This procedure can be technically demanding and associated with a wide range of adverse events. Technically failed ERCP may result in complications, need for additional procedures and their associated costs. Similar to EUS, ERCP is operator dependent and requires acquisition of certain technical and cognitive skills. There are limited data on learning curves and competence in ERCP, a cannulation rate of >80% (with some suggesting >90%) has been considered a surrogate for trainee competency. The American Society of Gastrointestinal Endoscopy (ASGE) recommends a minimum of 180 total procedures, the majority of which are therapeutic before competency can be achieved. However, this threshold is based predominantly on biliary cannulation success rate and does not take into account procedure complexity and the different rates at which people learn. It is also important to note that none of the previous studies have evaluated learning curves and competency in other quality indicators such as successful stone extraction, traversing and dilating a stricture, stent placement to name a few.

Competency assessment tools: Previous competency assessment tools have focused primarily on a limited number of motor skills involved in EUS and ERCP with no procedure-related cognitive skill assessment. The investigators have designed a prospective comprehensive competency assessment tool using validated benchmarks to define competency thresholds. The EUS and ERCP Skills Assessment Tool (TEESAT) can be used in a continuous fashion throughout the duration of training to grade technical and cognitive skills in EUS and ERCP in a balanced manner.

Significance, Innovation and Impact on Training and Education With the launch of the ACGME's NAS, advanced endoscopy training programs should utilize competency based medical education and demonstrate that advanced endoscopy trainees (AETs) have attained the technical and cognitive skills required for safe and effective unsupervised practice in advanced endoscopy. Based on the investigators research, the investigators can draw two conclusions: a) individuals in training in any technical procedure acquire skills at different rates and emphasis needs to be shifted away from the number of procedures performed to performance metrics with defined and validated competency thresholds of performance and b) current guidelines of performing 150 EUS and 180 ERCPs are inadequate to achieve competence in EUS and ERCP, respectively. With the expanding indications and applications of EUS and ERCP and establishment of a number of "third tier" training programs in advanced endoscopy, standardization of the performance of EUS and ERCP and definition of competence and training among AETs is of paramount importance. The potential impacts of this study's results are multifold: i) facilitate the ability of training programs to evolve with the new ACGME/NAS reporting requirements, (ii) help program directors/trainers and trainees identify specific skill deficiencies in training and allowing for tailored, individualized remediation, (iii) create a centralized national database that would allow generation of "on-demand" detailed reports on how individual trainees are progressing compared with their peers across the nation, (iv) establish reliable and generalizable standardized learning curves (milestones) and competency benchmarks that national GI societies and training programs can use to develop credentialing guidelines.

APPROACH AND RESEARCH STRATEGY Setting and Subject Recruitment: Program directors and AETs at all advanced endoscopy programs registered with the ASGE will be invited to participate in this study and will be considered as study participants. AETs will complete a questionnaire to determine baseline characteristics and prior experience with EUS and ERCP. AETs' prior experience with EUS and ERCP will not be an exclusion criterion for this study.

Competency-assessment tool: TEESAT, a tool designed for competency assessment, will be used in a continuous fashion throughout the duration of training to grade technical and cognitive skills in EUS and ERCP. The investigators have demonstrated he feasibility and validity of this tool in previous studies.3-5 This tool uses a 4-point scoring system: 1-no assistance, 2-achieves with minimal verbal cues, 3-multiple verbal cues or hands on assistance needed, 4-unable to complete. Setting these anchors for specifics skills and behaviors for what is expected to achieve each score will ensure that the data collected are reproducible from one evaluator to the next. Technical aspects during EUS exams include grading of individual EUS stations and technical success in EUS-FNA. Cognitive aspects include identification of lesion of interest, appropriate classification of malignant tumors (TNM) staging characterization of subepithelial lesions. Technical aspects during biliary/pancreatic ERCP include endpoints such as intubation, achieving the short position, identification of the papilla, cannulation of desired duct, sphincterotomy, stone removal and stent placement. Cognitive aspects will include clear demonstration of indication of the procedure, appropriate use of fluoroscopy and logical plan based on cholangiogram/pancreatogram findings. This tool includes documentation of immediate and post-procedure complications. Grading protocol: All AETs will be introduced to both the cognitive and technical aspects of EUS and ERCP procedures at the onset of training. Although TEESAT is self-explanatory, the program directors at each center will ensure that the AETs and trainers are familiar with TEESAT's specific assessment parameters and score explanations. After completion of 25 hands-on EUS and ERCP exams, AETs will be graded on every ERCP and 3rd EUS exam by attending endoscopists (trainers) at each center. This frequency of grading was chosen based on the investigators pilot data. Grading of every 3rd EUS exam as opposed to every exam was chosen given the fairly homogenous population undergoing EUS compared to ERCP. Procedures that the AETs have no hands-on participation will be excluded for grading. If the exam eligible for grading is an incomplete procedure for reasons such as medical instability, this exam will not be used for grading. Trainers will complete the assessment immediately after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Program directors and AETs at all advanced endoscopy programs registered with the ASGE will be invited to participate in this study and will be considered as study participants.

Exclusion Criteria:

* N/A

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Program directors and AETs at all advanced endoscopy programs registered with the ASGE will be invited to participate in this study and will be considered as study participants.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Overall competency | Up to 12 months
  The proportion of advanced endoscopy trainees (AETs) that achieve overall competency in EUS and ERCP using a standardized competency assessment tool with a comprehensive data collection and reporting system.

SECONDARY OUTCOMES:
Competency in EUS | Up to 12 months
  The proportion of AETs that achieve competency in individual technical (EUS stations, and FNA) and cognitive (TMN staging) aspects of EUS.
Competency in ERCP | Up to 12 months
  The proportion of trainees that achieve competency in individual technical (cannulation rate, stone removal and stent placement) and cognitive (proficient use of cholangiography) aspects of ERCP.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver